CLINICAL TRIAL: NCT05095337
Title: A Phase I Mass Balance and Biotransformation Study of [14C]SHR1459 in Chinese Healthy Adult Male Volunteers
Brief Title: Study to Evaluate the Mass Balance and Biotransformation of [14C]SHR1459 in Healthy Adult Male Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SHR1459-I-108
Record Dates: First submitted 2021-03-01; First posted 2021-10-27 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Healthy Adult Male Volunteers

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [14C]SHR1459 (Experimental)
  Interventions: Drug: [14C]SHR1459

INTERVENTIONS:
Drug: [14C]SHR1459 — Patients will receive single dose of orally [14C]SHR1459 on Day 1.

SUMMARY:
Evaluate the Mass Balance and Biotransformation of [14C]SHR1459 in Healthy Adult Male Volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Signing the informed consent forms;
2. Healthy adult males;
3. Age: 18 Years to 45 Years(Including the boundary value);
4. Weight: Body mass index(BMI) between 19 and 26 kg/m2(Including the boundary value);

Exclusion Criteria:

Candidates who meet any of the following conditions will not be selected:

Laboratory examination:

1. Complete physical examination, laboratory examination (blood routine, blood biochemistry, urine routine, coagulation function, fecal occulted blood, thyroid function (FT3, FT4, TSH), 12-lead electrocardiogram, X-chest X-ray (orthostatic position), abdominal B-ultrasound (liver, bile, pancreas, spleen, kidney) and other abnormal and clinically significant examinations;
2. Ophthalmologic examination (slit lamp, intraocular pressure and fundus photography) with abnormal clinical significance;
3. Hepatitis B surface antigen or E antigen, hepatitis C antibody, HIV antibody and syphilis antibody, any of which are positive.

   Medical history:
4. Screening for use of any clinical trial drug within the first 3 months or withdrawal time shorter than the 6 half-life period of the trial drug at enrollment, whichever is the longest of the two;
5. CYP3A4 and CYP2C9 inducers or inhibitors were taken within 28 days before screening, as shown in Appendix 1.
6. Use of any prescription or over-the-counter drug, any vitamin product, health care drug or Chinese herbal medicine within 14 days prior to screening;

   Medical history and treatment history:
7. clinical symptoms or diseases of the heart that cannot be well controlled, such as :(1) heart failure of NYHA2 or above; (2) unstable angina pectoris; (3) myocardial infarction within 1 year; (4) supraventral or ventricular arrhythmia with clinical significance that requires treatment or intervention; (5) QTcF>450ms(male) at screening stage; (5) QTcF>450ms.
8. Patients who had undergone major surgery or whose surgical incision was not completely healed within 6 months before the screening period;Major surgery includes, but is not limited to, any surgery with a significant risk of bleeding, prolonged general anesthesia, or an open biopsy or significant traumatic injury;
9. Screening for abdominal fistula, gastrointestinal perforation or abdominal abscess in the first 6 months;
10. Screening for clinically significant bleeding symptoms or definite bleeding tendency, such as gastrointestinal bleeding and bleeding ulcer, in the first 3 months;
11. Hemorrhoids or perianal diseases with regular/bleeding in the stool;Patients with gastrointestinal dysfunction, such as irritable bowel syndrome and inflammatory bowel disease, may be affected by drug absorption as determined by researchers;
12. Allergic persons, including those with a history of severe drug allergy or drug allergy, and those with known allergy to SHR6390 or similar drugs and excipients;Allergic to any food ingredients or has special requirements on diet, cannot follow the unified diet;
13. A history of any clinically serious illness or condition, including but not limited to circulatory, endocrine, nervous, digestive, urinary, or blood, immune, mental, and metabolic diseases, that the investigator considers to be likely to affect the results of the study;

    Living Habits:
14. Habitual constipation or diarrhea;
15. Heavy drinking or regular drinking in the six months preceding the screening period, i.e. drinking more than 14 units of alcohol per week (1 unit =285 mL beer or 25 mL spirits of 40% alcohol or 100 mL wine);Or alcohol breath test results at screening period ≥20 mg/ dL;
16. Those who had smoked more than 5 cigarettes per day on average in the 3 months before the screening period or habitually used nicotine containing products and were unable to quit during the test period;
17. Substance abuse or use of soft drugs (e.g., marijuana) in the 3 months prior to the screening period or use of hard drugs (e.g., cocaine, amphetamines, phenylcyclohexidine, etc.) in the 1 year prior to the screening period;Or screening for positive urine drug abuse (drug) tests;
18. habitual consumption of grapefruit juice or excessive consumption of tea, coffee and/or caffeinated beverages and failure to abstain during the study period;

    Other:
19. Those with a history of fainting needle or blood, have difficulty in blood collection or cannot tolerate vein puncture for blood collection;
20. Workers engaged in conditions requiring long-term exposure to radioactivity;Or have significant radiation exposure (≥2 chest/abdomen CT, or ≥3 other types of X-ray examinations) within 1 year before the test or have participated in the radiopharmaceutical labeling test;

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2022-06-07 (Actual); Primary Completion 2022-07-05 (Estimated); Study Completion 2022-07-25 (Estimated)

PRIMARY OUTCOMES:
Tmax | up to Day 21 (approx) from the start of administration.
Cmax | up to Day 21 (approx) from the start of administration.
AUC0-t | up to Day 21 (approx) from the start of administration.
AUC0-∞ | up to Day 21 (approx) from the start of administration.
t1/2 | up to Day 21 (approx) from the start of administration.
CL/F | up to Day 21 (approx) from the start of administration.
Vz/F | up to Day 21 (approx) from the start of administration.
Total radioactivity ratio for blood/plasma | up to Day 21 (approx) from the start of administration.
cumulative recovery of total radioactive substances in urine and/or feces; | up to Day 21 (approx) from the start of administration.
Percentage of metabolites in urine and feces in dose administration (% of dose administration) or percentage of circulating metabolites in plasma in total exposure AUC (%AUC); | up to Day 21 (approx) from the start of administration.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events(AEs) and Serious Adverse Events. | up to Day 21 (approx) from the start of administration.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided